CLINICAL TRIAL: NCT02365350
Title: A Randomized, Controlled, Open Trial Comparing a 17 G Single Lumen Aspiration Needle With a Modified Double Lumen Needle System (STEINER-TAN Needle®) for Follicular Flushing During Oocyte Pick-up in IVF Patients With Poor Ovarian Response
Brief Title: Randomized Clinical Trial on Follicular Flushing in IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. M.Sc. Georg Griesinger, Prof. Dr. med. M.Sc. Georg Griesinger, University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-244
Record Dates: First submitted 2015-02-06; First posted 2015-02-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- STEINER-TAN Needle® (Experimental): All visible follicles regardless of size in both ovaries will be aspirated and flushed three times by the STEINER-TAN Needle.
  Interventions: Procedure: STEINER-TAN Needle®
- 17G single lumen needle (Active Comparator): In the control group all visible follicles regardless of size in both ovaries will be aspirated by the 17G single lumen needle.
  Interventions: Procedure: 17 G single lumen needle

INTERVENTIONS:
Procedure: STEINER-TAN Needle® — A purpose built new double lumen needle with little dead space.
  Arms: STEINER-TAN Needle®
Procedure: 17 G single lumen needle — A conventional single lumen IVF aspiration needle.
  Arms: 17G single lumen needle

SUMMARY:
The primary objective is to demonstrate superiority of follicle flushing with the STEINER-TAN Needle® as compared to single lumen aspiration in terms of numbers of COCs retrieved.

DETAILED DESCRIPTION:
Rationale:

Since the number of oocytes available for IVF is a determinant of the cumulative chance of a patient to achieve pregnancy, it is of paramount importance to optimize the number of oocytes at oocyte pick-up. This especially for a fraction of patients, who despite high-dosed FSH stimulation, produce only a small number of growing follicles (poor response).

Objective:

The primary objective is to demonstrate superiority of follicle flushing with the STEINER-TAN Needle® as compared to single lumen aspiration in terms of numbers of COCs retrieved.

The secondary objective is to study differences in numbers of mature oocytes, proportion of patients undergoing embryo transfer, pregnancy rate, duration of the procedure, impact on patient burden (as assessed by the DASS 21, the German pain questionnaire [www.dgss.org]) and subjective patient experience.

Study design:

Prospective, single-center, randomized controlled, open trial comparing a 17G single lumen aspiration needle with a modified double lumen needle system (STEINER-TAN Needle®) for follicular flushing during oocyte pick-up in IVF patients with poor ovarian response.

Study population:

Patients with a BMI < 35 kg/m2 and an indication for IVF or ICSI with or without ovarian stimulation presenting with ≤ 5 follicles >10mm in the ovaries at the end of the follicular phase of the treatment cycle will be eligible for inclusion. Final oocyte maturation is to be induced by hCG administration as soon as the leading follicle reaches a mean diameter of 18mm or the day thereafter.

Intervention:

Eighty (n=80) patients will be randomly allocated on the day when the decision is taken to administer hCG to one of the following two procedures. In the study group all visible follicles regardless of size in both ovaries will be first aspirated and then flushed at least three times by the STEINER-TAN Needle® system. In the control group all visible follicles regardless of size in both ovaries will be aspirated by the 17G single lumen needle.

Main study parameters/endpoints:

The main study parameter/endpoint is the mean number of COSs per patient randomized.

Secondary endpoints are the mean number of mature metaphase II oocytes per patient and per COC retrieved per patient, the number of fertilized (2PN) oocytes, the fertilization rate (number of 2PN oocytes/number of injected or inseminates oocytes), the pregnancy rate (viable pregnancy at 6-7 gestational weeks/randomized patient), the mean DASS 21 score after the procedure, the mean duration of the procedure (min, sec), the COC retrieval rate per puncture follicle and the proportion of randomized patients not reaching embryo transfer. Furthermore, the patients will be interviewed about their overall experience of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects undergoing IVF or ICSI treatment with or without ovarian stimulation
* ≤ 5 follicles >10 mm at the end of the follicular phase as assessed by transvaginal ultrasound
* Presence of two ovaries
* Willingness to participate
* Informed consent

Exclusion Criteria:

* BMI <18 or >35 kg/m2
* Ovaries cannot be reached (e.g. heterotopic ovaries)
* Age <18 or >45

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Mean number of COSs per patient randomized. | 1 day

SECONDARY OUTCOMES:
Mean number of mature metaphase II oocytes | 1 day
Pregnancy rate | 7 weeks
Mean number of fertilized (2PN) oocytes | 2 days
Mean DASS 21 score after the procedure | 1 day
Mean duration of the procedure. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Georg Griesinger, MD MSc PhD, Principal Investigator — University of Luebeck
Locations (1):
- Universitäres Kinderwunschzentrum Lübeck, Lübeck, Schleswig-Holstein, Germany